CLINICAL TRIAL: NCT03751189
Title: Trauma to Permanent Incisors and Overjet in Libyan Children
Brief Title: Role of Overjet and Trauma in Libyan Children
Status: Completed | Type: Observational
Sponsor: sudhir rama varma (Other)
Responsible Party: Sponsor-Investigator, sudhir rama varma, Assistant Professor, Ajman University
Organization: Ajman University (Other)
Other Study IDs: 07/16
Record Dates: First submitted 2018-11-18; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Trauma; Overjet
Keywords: trauma; overjet; libya; schoolchildren
MeSH Terms: conditions — Wounds and Injuries; Overbite

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Traumatic dental injuries are one of the commonly encountered dental emergencies. Missing anterior tooth in children due to any injury can be a source of considerable physical and psychological discomfort for the child. These consequences also have significant impact on parents, who are generally concerned with esthetic and economic aspects of this problem. It varies from small crack in the enamel to complete loss of the tooth. Injury to children teeth can be both painful and traumatic to the children

DETAILED DESCRIPTION:
Traumatic injuries to anterior teeth have reported by several investigators. In Asia and Africa, the prevalence of TDI to anterior teeth among adolescents ranges from 4% to 35% and 15% to 21%, respectively and in America and Europe, the prevalence varied from 15% to 23% and 23% to 35%, respectively . 50% of school children have sustained traumatic injuries prior to graduation . A contributing factors make children susceptible to injuries have been widely investigated. These factors included Class-II, div.1 malocclusion, increased overjet . 71% to 92% of all injuries sustained in a lifetime occur before the age of 19 years, which occur at home, followed by school and public places.The aim of this study is to assess the mean overjet value in Libyan children and to examine the relationship between increased overjet and trauma to permanent incisor teeth

ELIGIBILITY:
Inclusion Criteria:

* Libyan children.
* The permanent incisors are present & sufficiently erupted.

Exclusion Criteria:

* Non Libyan children.
* The permanent incisors are absent, or un-sufficiently erupted.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: . Total of 2015 Libyan school children aged 7 to 16 years from urban (Tobruk) and rural (Kufra) areas were examined in the main study. The children were of almost equal number of both sexes from each age group
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Number of school children with overjet | From baseline to 10 months
  Presence of overjet among school children, is evaluated by observational method,measured by 1-1mm-3mm;2-3mm-5mm;3-5mm<

SECONDARY OUTCOMES:
Dental trauma among school children | From baseline to 10 months
  Presence of trauma ,by observational method; Grading done by 0- No trauma;1-trauma related to incisal region;2-trauma related to mid half;3-trauma pertaining to cervical region

IPD SHARING:
Plan to Share IPD: Undecided